CLINICAL TRIAL: NCT06989346
Title: Impact of Perioperative Hyperoxia on Cancer Recurrence and Mortality After Elective Colorectal Cancer Surgery
Acronym: OncO2
Status: Completed | Type: Observational
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Sponsor
Other Study IDs: OncO2
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Recurrence; Survival Rate; Mortality; Colorectal Surgery; Hyperoxia
Keywords: Hyperoxia; Recurrence-free Survival; Colorectal Surgery
MeSH Terms: conditions — Recurrence; Hyperoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hyperoxia: Perioperative hyperoxia (FiO₂ > 0.8)
- Control: Conventional perioperative oxygen therapy (FiO₂ < 0.4)

SUMMARY:
The goal of this observational study is to evaluate whether perioperative hyperoxia (FiO₂ > 0.8), compared to conventional oxygen therapy (FiO₂ < 0.4), is associated with increased cancer recurrence and mortality in patients undergoing curative elective colorectal cancer surgery.

DETAILED DESCRIPTION:
In 2016, the World Health Organization (WHO) recommended the use of perioperative hyperoxia (FiO₂ > 0.8) to reduce the risk of postoperative surgical site infections (SSIs). However, the WHO also highlighted potential adverse effects associated with hyperoxia, including increased cancer recurrence and mortality. This study aims to evaluate whether perioperative hyperoxia (FiO₂ > 0.8), compared to conventional oxygen therapy (FiO₂ < 0.4), is associated with increased cancer recurrence and mortality in patients undergoing curative elective colorectal cancer surgery.

This study is a follow-up of a previously published cohort originally designed to assess whether FiO₂ > 0.8 was associated with a higher incidence of perioperative cardiovascular complications. In this follow-up, oncological recurrence and mortality events were recorded at least three years after the index surgery. The primary outcome was recurrence-free survival over the follow-up period, analyzed using Kaplan-Meier curves and a Cox proportional hazards model. The secondary outcome was the 3-year mortality rate, analyzed using the Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old;
* Scheduled for major elective colorectal surgery under general anaesthesia with tracheal intubation.

Exclusion Criteria:

* Non-oncologic surgery or non-curative oncological surgery
* Pregnant or breastfeeding women
* Chronic obstructive pulmonary disease (forced expiratory volume in one second <50% or in need of domiciliary oxygen thera-py)
* Acute coronary event or stroke during the previous six weeks (before the surgery)
* Chronic renal failure requiring renal replacement therapy;
* Predicted length of stay of less than one day;
* Any patient that has received general anaesthesia during the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with colorectal cancer, eligible for a scheduled colorectal surgery with a curative intention
Sampling Method: Non-Probability Sample
Enrollment: 403 (Actual)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Recurrence-free Survival | Follow-up period (at least 3 years since surgery)
  Length of time from the end of primary treatment (surgery in this case) until the evidence of cancer recurrence (locoregional or systemic) or death in the last follow-up

SECONDARY OUTCOMES:
Mortality | 3-year follow-up period
  Percentage of global mortality (not exclusively related to the oncologic disease)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sadurní, MD, Principal Investigator — Hospital del Mar; Laura Castelltort, MD, Study Director — Hospital del Mar
Locations (1):
- Hospital del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
We need to pursue additional conversations with our organization to request to share IPD.

REFERENCES:
- [Background] Sadurni M, Castelltort L, Rivera P, Gallart L, Pascual M, Duran X, Grocott MP. Perioperative hyperoxia and myocardial injury after surgery: a randomized controlled trial. Minerva Anestesiol. 2023 Jan-Feb;89(1-2):40-47. doi: 10.23736/S0375-9393.22.16634-4. Epub 2022 Oct 25. PMID 36282221
- [Background] Podolyak A, Sessler DI, Reiterer C, Fleischmann E, Akca O, Mascha EJ, Greif R, Kurz A. Perioperative Supplemental Oxygen Does Not Worsen Long-Term Mortality of Colorectal Surgery Patients. Anesth Analg. 2016 Jun;122(6):1907-11. doi: 10.1213/ANE.0000000000001316. PMID 27195634
- [Background] Meyhoff CS, Jorgensen LN, Wetterslev J, Siersma VD, Rasmussen LS; PROXI Trial Group. Risk of new or recurrent cancer after a high perioperative inspiratory oxygen fraction during abdominal surgery. Br J Anaesth. 2014 Jul;113 Suppl 1:i74-i81. doi: 10.1093/bja/aeu110. Epub 2014 May 23. PMID 24860156